CLINICAL TRIAL: NCT06442072
Title: Global Controlled Trial on Effects of a Guided Online Self-Help Program for of Ambitious Altruists on Their Mental Health, Wellbeing, and Productivity
Brief Title: Global Controlled Trial on Effects of an Online Self-Help Program for of Ambitious Altruists on Their Mental Health, Wellbeing, and Productivity: Comparing Versions With IFS vs. CBT, Buddy- vs. Group-, Standard- vs. Minimum-Guidance Intensity.
Acronym: CT_DoBetter
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rethink Wellbeing (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CT2024RW
Record Dates: First submitted 2024-05-18; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Treatment Adherence and Compliance; Anxiety; Depression; Mental Health Issue; Quality of Life; Well-Being, Psychological; Social Functioning; Cognitive Dysfunction; Interpersonal Relations; Self Esteem; Loneliness; Functioning, Psychosocial; Functioning, Social
Keywords: Mental Health; CBT; Productivtiy; Controlled trial; Effectiveness; Prevention; guided self-help; IFS
MeSH Terms: conditions — Treatment Adherence and Compliance; Anxiety Disorders; Depression; Psychological Well-Being; Social Adjustment; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CBT Group Standard Guidance (Active Comparator): * 9 group sessions, at week 0-6, 8, 12, 18
  * groups of 4-6 peers and a trained facilitator
  * participants work through the tailored Third Wave CBT workbook by Rethink Wellbeing, one chapter each week
  * in between sessions, people practice the new skills learned in the workbook and are supported in an online community, guided by a trained psychologist and psychotherapist
  Interventions: Behavioral: guided online self-help program
- CBT Buddy Standard Guidance (Active Comparator): * 9 1:1 sessions after buddies get training in supporting each other - at week 0-6, 8, 12, 18
  * groups of up to 30 peers and a trained facilitator
  * participants work through the tailored Third Wave CBT workbook by Rethink Wellbeing, one chapter each week
  * in between buddy-sessions, people practice the new skills learned in the workbook and are supported in an online community, guided by a trained psychologist and psychotherapist
  Interventions: Behavioral: guided online self-help program
- CBT Group Minimum Guidance (Active Comparator): * 3 instead of 9 sessions, in week 1, 8 and 16.
  * groups of up to 30 peers and a trained facilitator
  * participants work through the tailored Third Wave CBT workbook by Rethink Wellbeing, one chapter each week
  * in between, people practice the new skills learned in the workbook and are supported in an online community, guided by a trained psychologist and psychotherapist
  Interventions: Behavioral: guided online self-help program
- IFS Group Standard Guidance (Active Comparator): * 9 group sessions, at week 0-6, 8, 12, 18
  * groups of 4-6 peers and a trained facilitator
  * Internal Family Systems methods taught instead of CBT methods as in every other group
  * participants work through the book "Self-Therapy: A Step-By-Step Guide to Creating Wholeness and Healing Your Inner Child Using IFS, A New, Cutting-Edge Psychotherapy" by Jay Earley, a few chapters each week
  * in between, people practice the new skills learned in the workbook and are supported in an online community, guided by a trained psychologist and psychotherapist
  Interventions: Behavioral: guided online self-help program

INTERVENTIONS:
Behavioral: guided online self-help program — 16 weeks of training and application of psychotherapeutic methods

SUMMARY:
This study aims to compare different versions of a 16-week online self-help program in terms of their effect on self-assessed mental health, well-being, and productivity. The versions differ in their intensity (standard, low) and type (buddy, group) of guidance, the applied psychotherapeutic approaches taught (IFS, CBT). We expect to recruit a sample of ~150 ambitious altruists and have them self-select into the four program versions. Participants take part in surveys before, at weeks 8, 12, and 16 to self-assess their productivity, mental health burden, quality of life, and other risk and protection factors. Weekly screenings will provide data on objective and subjective success components such as participant engagement, working alliance, and treatment adherence, which will be correlated with primary and secondary outcomes.

DETAILED DESCRIPTION:
Aim:

This study aims to compare different versions of an online self-help program in terms of their effect on self-assessed mental health, well-being, and productivity. The goal is to find out if a version might be more effective or similarly effective but less costly than the original one.

Control groups:

The original program version is an 8-week course with weekly guided group sessions of 2 hours: Third Wave CBT methods are taught by a workbook and practised in between the sessions. The pre-post results, on 42 ambitious altruists, showed significant moderate effects on all scales after week 12. In this study, we aim to compare the effects of the original version with 1. one using a buddy instead of the group format, 2. one using less guidance (3 instead of 9 group sessions), and 3. one using Internal Family Systems instead of Third Wave CBT. Instead of 8 weeks, we spaced out the same amount of sessions for the program after week 6, so that the last follow-up session will take place for everyone at week 16 now.

Sample:

We expect to deliver the program to ~150 participants, and each version to at least 25 of those. Ambitious altruists will be recruited via posts on Facebook and Slack online groups and personal contact to organizations associated with Effective Altruism. People will self-select into the different program versions. We exclude those in acute crisis, those with very low self-assessed social competence, and those who report not being ambitiously altruistic. We match groups and buddies based on availability and on, who we believe will bond better, i.e., similar age and career stage.

Measurements. Participants take part in Google form surveys before, at weeks 8, 12, and 16. These measure productivity (WPAI:GH), mental health burden (symptoms of interpersonal sensitivity, and OCD by BSI, depressiveness and anxiety by GAD7 & PHQ8), quality of life (WHOQOL-BREF, MHC-SF, ONS-4 LS), and other relevant factors (loneliness by UCLA-3, self-esteem by Rosenberg Self-esteem Scale, connection/will to do good by IWAH). An independent researcher, likely from Maastricht University, will likely check our data, calculate the results, and publish a paper about it to reduce potential biases. Also, participants' engagement will be assessed, i.e., no-shows, and dropouts, and participants attend a weekly screening in weeks 1-8, 12, and 16 to rate different success components, e.g. session engagement, working alliance, and treatment adherence. Those measures will be correlated with the primary and secondary outcomes at one point to see what influences outcomes and how strongly.

We applied to get an official letter of exemption from an ethics review due to these reasons:

* The study is only part of the already existing programs, nothing is changed in the operations affecting the participants due to the evaluation/study run
* Measurements are part of routine progress tracking
* The data is being used for publication purposes but does not introduce new risks
* The interventions as well as the data collection are 100% non-invasive and include a signed participant consent.
* The sampling excludes potentially vulnerable individuals, i.e., those in a current crisis.

ELIGIBILITY:
Exclusion Criteria:

* average of self-assessed sociality negative
* people in acute crisis (they confirm and sign to not be in such a state)
* people who self-report not to be ambitiously altruistic, i.g., not involved in the effective altruism community, or working on or planning to work on something impactful that might help others.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Productivity | Week 0, 8, 12, 16
  by WPAI:GH: Work Productivity & Activity Impairment Questionnaire. The item values will be merged into one scale by turning each into a z-score while higher numbers will mean a higher productivity, and then calculating the average.
Mental health burden | Week 0, 8, 12, 16
  symptoms of interpersonal sensitivity, and executive dysfunction by BSI, of depressiveness and anxiety by GAD7 & PHQ8. The scores will be merged into one by turning each of the 4 scales into a z-score while higher numbers will mean a larger burden, and then calculating the average.
Wellbeing | Week 0, 8, 12, 16
  psychological, social and emotional functioning as well as quality of life by WHOQOL-BREF, MHC-SF ONS-4 LS. The scores will be merged into one by turning each of the scales into a z-score while higher numbers will mean a higher wellbeing, and then calculating the average.

SECONDARY OUTCOMES:
Loneliness | Week 0, 8, 12, 16
  UCLA-3
Self-esteem | Week 0, 8, 12, 16
  Rosenberg Self-esteem Scale
Connection/will to do good | Week 0, 8, 12, 16
  by IWAH
Program dropout | Week 0, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16
  % of participants announcing their drop-out or not showing up to 2+ sessions, higher numbers mean higher dropout
Weekly engagement | Week 1, 2, 3, 4, 5, 6, 8, 12, 16
  Treatment adherence, session engagement, working alliance, session attendance rate. The scores will be merged into one by turning each of the values into a z-score while higher numbers will mean a higher engagement, and then calculating the average.

CONTACTS AND LOCATIONS:
Overall Officials: Inga Grossmann, PhD., Study Director — Rethink Wellbeing
Locations (1):
- Rethink Wellbeing, Wapenveld, Netherlands

IPD SHARING:
Plan to Share IPD: No